CLINICAL TRIAL: NCT07119593
Title: Boosting Myocardial Preconditioning With High-Intensity Intradialytic Exercise: A Preliminary Study
Brief Title: Exercise Intensity
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Chris McIntyre, Nephrologist, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 15956
Record Dates: First submitted 2025-06-19; First posted 2025-08-13 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Dialysis; Cardioprotection

STUDY DESIGN:
Intervention Model Description: Open label, randomized, controlled, crossover trial with 3 conditions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Randomization Order 1 (Other): Participants will be randomized into one of the three conditions indicating the order in which they will receive the exercise intervention. Randomization Order 1 will receive control (no exercise) week one. Week 2 the participant will have a moderate intensity exercise treatment and week three the participant will have a high intensity exercise treatment. All sessions (i.e. HD-Cont, HD-Mod and HD-High) will be performed on one of the patient's three days of weekly dialysis. Each patient will consistently perform all sessions on the same day of dialysis throughout the study. The three sessions will be separate by at least one week to avoid potential carryover effects.
  Interventions: Other: Intradialytic Cycling
- Randomization Order 2 (Experimental): Participants will be randomized into one of the three conditions indicating the order in which they will receive the exercise intervention. Randomization Order 2 will receive moderate intensity exercise week one. Week 2 the participant will have high intensity exercise and week three the participant will have control (no exercise). All sessions (i.e. HD-Cont, HD-Mod and HD-High) will be performed on one of the patient's three days of weekly dialysis. Each patient will consistently perform all sessions on the same day of dialysis throughout the study. The three sessions will be separate by at least one week to avoid potential carryover effects.
  Interventions: Other: Intradialytic Cycling
- Randomization 3 (Experimental): Participants will be randomized into one of the three conditions indicating the order in which they will receive the exercise intervention. Randomization Order 3 will receive high intensity exercise week one. Week 2 the participant will have control (no exercise) and week three the participant will have a moderate intensity exercise treatment. All sessions (i.e. HD-Cont, HD-Mod and HD-High) will be performed on one of the patient's three days of weekly dialysis. Each patient will consistently perform all sessions on the same day of dialysis throughout the study. The three sessions will be separate by at least one week to avoid potential carryover effects.
  Interventions: Other: Intradialytic Cycling

INTERVENTIONS:
Other: Intradialytic Cycling — Intradialytic exercise has emerged as a safe and effective non-drug therapeutic approach to improve cardiovascular health and is now recommended for people undergoing hemodialysis treatment. Administration of a higher intensity exercise could offer better cardio-protective mechanisms and if the efficacy of cardiovascular protection is proven, it could be developed as a therapeutic option in the dialysis population.

SUMMARY:
Patients receiving regular hemodialysis (HD) treatments are at a higher risk of cardiovascular events and death as HD can cause a decrease in the pumping of the heart during treatment called 'stunning'. Intradialytic exercise has emerged as a safe and effective non-drug approach to improve cardiovascular health and is now recommended for patients undergoing HD. It is currently advised that HD patients engage in at least 30 minutes of moderate to vigorous exercise three times per week. This study will evaluate the impact of exercise intensity in the HD population and determine if high impact exercise can offer better protection to the heart against HD-induced myocardial stunning.

DETAILED DESCRIPTION:
This will be the first randomized, cross-controlled trial evaluating the impact of exercise intensity in the HD population. If the efficacy of cardiovascular protection is proven, it could be developed as a therapeutic option in the dialysis population.

ELIGIBILITY:
Inclusion Criteria:

* Must be on chronic hemodialysis for at least 3 months
* Age ≥ 18 years of age
* Willing and able to provide informed consent

Exclusion Criteria:

* Regular vigorous exercise outside hemodialysis
* > 79 years of age
* Intradialytic exercise in the past 3 months
* Poor echogenicity
* Acute coronary syndrome in the past 3 months
* Unstable arrhythmia/angina
* Shortness of breath at rest or with minimal activity
* Symptomatic hypoglycemia (>2x/week in the week prior to enrolment)
* Symptomatic peripheral arterial disease
* Unable or deemed unsafe to exercise for any reason
* Severe musculoskeletal or orthopedic conditions
* Aortic stenosis
* Hypertrophic cardiopathy
* Severe pulmonary hypertension
* Symptomatic hypertension

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-09-22 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in the number of left ventricular segments undergoing a greater than 20% reduction in longitudinal strain as detected by echocardiogram. | Week 1 to Week 3
  An echocardiogram will be completed pre-hemodialysis (HD) treatment and at peak hemodynamic stress (30 minutes before the end of HD treatment) at each of the study sessions. Images will be captured in the left lateral position and standard apical 4, and 2 chamber views will be recorded for analysis using automated speckle-training software. (EchoPac, GE Healthcare)

SECONDARY OUTCOMES:
Evaluate potential targets of exercise induced cardio protection by evaluating their effects on endothelial function. | Week 1 to Week 3
  Endothelial function will be assessed by measuring the dilatory response of the brachial artery to increased blood flow generated by reactive hyperemia in the downstream forearm. At each study session participants are placed in the supine position and the brachial artery of the non-dominant arm, or the non-distended arm is scanned in longitudinal section using a 12 MHz linear transducer connected to a Vivid Q echograph (GE, /USA) supplemented by an electrocardiogram (ECG).
Evaluate whether the increase in exercise intensity leads to a differential modulation of potential cardioprotective mechanisms, by evaluating their effects on hemodynamic responses (Blood Pressure) | Week 1 to week 3
  Systolic blood pressure (SBP), Diastolic blood pressure (DBP) and mean arterial pressure (MAP) will be measured using an automated blood pressure monitor integrated into the dialysis machine. Values will be monitored throughout each study visit.
Evaluate whether the increase in exercise intensity leads to a differential modulation of potential cardioprotective mechanisms, by evaluating their effects on hemodynamic responses (CV Insight Monitoring) | Week 1 to Week 3
  The CV Insight contact device is non-invasive continuous hemodynamic real time monitoring system use to assess cardiovascular and respiratory status using percutaneous photoplethysmography. The device will be attached to the right of the patient's forehead midline., approximately 2.5cm above the level of the nose pre-dialysis and will remain intact until the patient is disconnected from the dialysis machine at each study session. Once attached, baseline recording will be obtained, and hemodynamic data will continuously be captured.
Evaluate whether the increase in exercise intensity leads to a differential modulation of potential cardioprotective mechanisms, by evaluating their effects on hemodynamic responses (Finapres) | Week 1 to Week 3
  The Finometer utilizes a finger-cuff method to detect beat-to-beat changes in digital arterial diameter using an infrared photoplethysmography. The time averaged data is subsequently downloaded to a computer-based analysis program for analysis. The finger-cuff will be placed on the participant's index finger at each study visit and will remain in place through the entirety of the visit.
Evaluate whether the increase in exercise intensity leads to a differential modulation of potential cardioprotective mechanisms, focusing on blood markers. | Week 1 to Week 3
  Blood samples will be collected from the participants dialysis access before HD and at peak stress at each study visit for biochemistry, proteomic analysis and translational approach.

CONTACTS AND LOCATIONS:
Overall Officials: Chris McIntyre, MBBS DM, Principal Investigator — London Health Sciences Centre
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Not Yet Determined
Supporting Information: Study Protocol
Time Frame: Not Yet Determined
Access Criteria: Not Yet Determined